CLINICAL TRIAL: NCT01029795
Title: A 12-Week, Phase 2, Randomized, Double-Blind, Active-Controlled Study of LY2599506 Given as Monotherapy or in Combination With Metformin in Patients With Type 2 Diabetes Mellitus
Brief Title: A Study of LY2599506 (Oral Agent Medication: Glucokinase Activator 1) in Type 2 Diabetes Mellitus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to nonclinical safety findings
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13272; I2Q-MC-GMAJ (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-12-09; First posted 2009-12-10 (Estimated); Results first posted 2011-10-26 (Estimated); Last update posted 2011-12-02 (Estimated); Status verified 2011-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Glyburide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY2599506 (Experimental): Combinations of 50-milligram (mg) or 100-mg capsules of LY2599506 or matching placebo capsules (each dose contains at least 1 capsule of active drug). LY2599506 will be administered, based on predefined glycemic targets, in escalating doses from 100 mg/day up to 800 mg/day.
  Interventions: Drug: LY2599506; Drug: Placebo
- Glyburide (Active Comparator): Combinations of 2.5-mg capsules of Glyburide or matching placebo capsules (each dose contains at least 1 capsule of active drug). Glyburide will be administered, based on predefined glycemic targets, in escalating doses from 5 mg/day up to 20 mg/day.
  Interventions: Drug: Glyburide; Drug: Placebo

INTERVENTIONS:
Drug: LY2599506 — Administered orally (po), twice daily (BID) prior to morning and evening meals for 12 weeks
  Other Names: Glucokinase Activator 1
  Arms: LY2599506
Drug: Glyburide — Administered po, BID daily prior to morning and evening meals for 12 weeks
  Arms: Glyburide
Drug: Placebo — Matching placebo capsules administered po, BID prior to morning and evening meals for 12 weeks

SUMMARY:
The purpose of this study is to help answer the following research question(s):

* To test if taking LY2599506 for 12 weeks controls blood sugar better than taking glyburide for 12 weeks.
* To evaluate the safety of LY2599506 in participants with diabetes.
* To determine if LY2599506 has the ability to control blood sugar in participants with diabetes.
* To determine how much LY2599506 should be given to participants.
* To determine if LY2599506 has an effect on a participant's weight.

The study design consists of 4 study periods: a screening period, a 4-week dose adjustment period, an 8-week treatment period, and a 4-week follow up period.

ELIGIBILITY:
Inclusion Criteria:

* Have type 2 diabetes mellitus prior to entering the trial
* Are currently being treated with diet and exercise therapy consistent with the local standards of medical care
* Treated with: Diet and exercise alone; or Diet and exercise in combination with a stable dose of metformin for at least 3 months prior to entering the trial; or Diet and exercise in combination with a stable dose of sulfonylurea for at least 3 months prior to entering the trial; or Diet and exercise in combination with stable doses of metformin and sulfonylurea for at least 3 months prior to entering the trial and have had diabetes for at least 6 years.
* Have an HbA1c value between 7% and 10%
* Are women not of child-bearing potential due to surgical sterilization (hysterectomy or bilateral oophorectomy or tubal ligation) or menopause. Male patients will be advised to use a reliable method of birth control during the study and until 3 months after the last dose of study medication if their partner is of child-bearing potential.

Exclusion Criteria:

* Use of insulin or any antidiabetic agent other than metformin or sulfonylurea during the 3 months prior to entering the trial.
* Have a gastrointestinal disease that significantly impacts gastric emptying or motility (for example, severe gastroparesis or pyloric stenosis), in the opinion of the Investigator, or have undergone gastric bypass or gastric banding surgery.
* Have had more than 1 episode of severe hypoglycemia within 6 months prior to entry into the study, or are currently diagnosed as having hypoglycemia unawareness
* Have had 2 or more emergency room visits or hospitalizations due to poor glucose control in the past 6 months.
* Have cardiac autonomic neuropathy (for example, resting tachycardia or orthostatic hypotension), based on clinical signs, symptoms, or appropriate diagnostic testing.
* Have cardiac disease with functional status that is New York Heart Association Class II, III, or IV or a history of myocardial infarction, unstable angina, or decompensated congestive heart failure in the past 6 months.
* Have poorly controlled hypertension (that is, mean systolic blood pressure >160 mm Hg or mean diastolic blood pressure >100 mm Hg) history of malignant hypertension, evidence of renal artery stenosis, and/or evidence of labile blood pressure including symptomatic postural hypotension. Doses of antihypertensive medications must be stable for 30 days before randomization.
* Have fed or fasting state hypertriglyceridemia (defined as >6.8 millimoles per liter [mmol/L], 600 milligrams per deciliter [mg/dL]) at screening. If taking lipid-lowering agents, doses of these medications must be stable for 30 days prior to randomization.
* Have obvious clinical signs or symptoms of liver disease, acute or chronic hepatitis, or repeated alanine transaminase (ALT) levels >2.5 times the upper limit of the reference range at screening.
* Have evidence of a significant active, uncontrolled endocrine or autoimmune abnormality, as judged by the Investigator at screening.
* Have an active or untreated malignancy or have been in remission from a clinically significant malignancy (other than basal or squamous cell skin cancer, in situ carcinomas of the cervix, or in situ prostate cancer) for less than 5 years.
* Have a history of seizure disorder.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-02; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9AM - 5PM Eastern Time (UTC/GMT - 5hours, EST), Study Director — Eli Lilly and Company
Locations (16):
- Australia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Elizabeth Vale, South Australia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., East Ringwood, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelberg, Victoria
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vienna, Austria
- Czechia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Holešov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prague
- Germany (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mainz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Neuss
- Israel (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jerusalem
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nahariya
- Russia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rostov-on-Don
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
- Spain (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Córdoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dos Hermanas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Teruel

RESULTS

PARTICIPANT FLOW:
Groups:
- LY2599506: Participants received up to 4 capsules by mouth (po), twice daily (BID), in combinations of 50 milligram (mg) or 100 mg capsules of LY2599506 or matching placebo capsules. (Each dose contained at least 1 capsule of active drug.) LY2599506 was administered, based on predefined glycemic targets, in escalating doses from 100 mg/day up to 800 mg/day.
- Glyburide: Participants received up to 4 capsules po BID in combinations of 2.5-mg capsules of Glyburide or matching placebo capsules. (Each dose contained at least 1 capsule of active drug.) Glyburide was administered, based on predefined glycemic targets, in escalating doses from 5 mg/day up to 20 mg/day.
Period: Overall Study
Arm/Group | LY2599506 | Glyburide
Started | 16 | 22
Completed | 0 | 0
Not Completed | 16 | 22
Not completed — Entry Criteria Not Met | 2 | 1
Not completed — Physician Decision | 2 | 1
Not completed — Sponsor Decision | 11 | 17
Not completed — Withdrawal by Subject | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LY2599506 | Glyburide | Total
Number analyzed (Participants) | 16 | 22 | 38
Age Continuous [Mean (Standard Deviation); unit: years] | 59.76 (6.74) | 59.38 (5.86) | 59.54 (6.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 10 | 15 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 16 | 21 | 37
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — There were no participants from Germany.
  participants
    Australia | 5 | 9 | 14
    Austria | 2 | 3 | 5
    Czech Republic | 1 | 2 | 3
    Israel | 2 | 1 | 3
    Russian Federation | 2 | 2 | 4
    Spain | 4 | 5 | 9
Duration of Diabetes in Years [Mean (Standard Deviation); unit: year] | 6.08 (5.03) | 7.73 (5.64) | 7.03 (5.38)
Percentage of Glycosylated Fraction of Hemoglobin A1c [Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin] — HbA1c: hemoglobin A1c, glycosylated fraction of hemoglobin A (%)
  percentage of glycosylated hemoglobin | 7.90 (0.75) | 7.78 (1.02) | 7.83 (0.91)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin A1c (HbA1c) at 12 Weeks
Description: Change in HbA1c from baseline following 12 weeks of therapy (HbA1c at week 12 minus HbA1c at baseline). Study GMAJ was terminated after enrolling 38 participants. Given the small sample size overall and per treatment arm, numerical summaries and statistical comparisons are not appropriate and may be scientifically/clinically misleading; therefore, this outcome measure is not presented.
Time Frame: Baseline, 12 weeks
Population: Data were reviewed but are not presented due to insufficient sample size.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | LY2599506 | Glyburide
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change From Baseline in the QT Interval in Electrocardiogram (ECG) at 12 Weeks and 16 Weeks
Description: Measures the QT interval in the ECG. Study GMAJ was terminated after enrolling 38 participants. Given the small sample size overall and per treatment arm, numerical summaries and statistical comparisons are not appropriate and may be scientifically/clinically misleading; therefore, this outcome measure was not analyzed.
Time Frame: Baseline, 12 weeks, 16 weeks
Population: The QT interval was not analyzed due to insufficient sample size.
Measure: Mean (Standard Deviation); unit: milliseconds (ms)
Arm/Group | LY2599506 | Glyburide
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change From Baseline in the Homeostasis Model Assessment (HOMA2) Pancreatic Beta Cell Function (%B) at 12 Weeks and 16 Weeks
Description: HOMA2 is a computer model that uses fasting plasma insulin and glucose concentrations to estimate steady state pancreatic beta cell function (%B) as a percentage of a normal reference population (normal young adults). The normal reference population was set at 100%. Study GMAJ was terminated after enrolling 38 participants. Given the small sample size overall and per treatment arm, numerical summaries and statistical comparisons are not appropriate and may be scientifically/clinically misleading; therefore, this outcome measure was not calculated or analyzed.
Time Frame: Baseline, 12 weeks, 16 weeks
Population: HOMA2 (%B) was not calculated due to insufficient sample size.
Measure: Mean (Standard Deviation); unit: percentage of beta cell function (%B)
Arm/Group | LY2599506 | Glyburide
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change From Baseline in the Homeostasis Model Assessment (HOMA2) of Insulin Sensitivity (%S) at 12 Weeks and 16 Weeks
Description: HOMA2 is a computer model that uses fasting plasma insulin and glucose concentrations to estimate insulin sensitivity (%S), as percentages of a normal reference population (normal young adults). The normal reference population was set at 100%. Study GMAJ was terminated after enrolling 38 participants. Given the small sample size overall and per treatment arm, numerical summaries and statistical comparisons are not appropriate and may be scientifically/clinically misleading; therefore, this outcome measure was not calculated or analyzed.
Time Frame: Baseline, 12 weeks, 16 weeks
Population: HOMA2 (%S) was not calculated due to insufficient sample size.
Measure: Mean (Standard Deviation); unit: percentage of insulin sensitivity (%S)
Arm/Group | LY2599506 | Glyburide
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change From Baseline in Triglycerides, Low-density Lipoprotein Cholesterol (LDL-C), High-density Lipoprotein Cholesterol (HDL-C), Non-HDL-C, Total Cholesterol, and Free Fatty Acids at 12 Weeks and 16 Weeks
Description: Fasting lipids were measured after an overnight fast. Lipids measured included triglycerides, HDL-C, LDL-C, non-HDL-C, total cholesterol, and free fatty acids. Study GMAJ was terminated after enrolling 38 participants. Given the small sample size overall and per treatment arm, numerical summaries and statistical comparisons are not appropriate and may be scientifically/clinically misleading; therefore, this outcome measure is not presented.
Time Frame: Baseline, 12 weeks, 16 weeks
Population: Data were reviewed but not presented due to insufficient sample size.
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | LY2599506 | Glyburide
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change From Baseline in the European Quality of Life -5 Dimension (EQ-5D) at 12 Weeks and 16 Weeks
Description: Assesses 5 health domains: mobility, self-care, usual activity, pain, and anxiety/depression with 3 options each. Total scores range from 5 (no problem) to 15 (more severe or frequent problems). An algorithm maps the 5 domain outcomes to a single index (0-1). A higher score indicates better perceived health state. Study GMAJ was terminated after enrolling 38 participants. Given the small sample size overall and per treatment arm, numerical summaries and statistical comparisons are not appropriate and may be scientifically/clinically misleading; therefore, this outcome measure was not analyzed.
Time Frame: Baseline, 12 weeks, 16 weeks
Population: Quality of life data were not analyzed due to insufficient sample size.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LY2599506 | Glyburide
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change From Baseline in the Diabetes Treatment Satisfaction Questionnaire (DTSQ) at 12 Weeks and 16 Weeks
Description: DTSQ, an 8-item questionnaire, measures satisfaction with treatment, perceived frequency of hyperglycemia, and perceived frequency of hypoglycemia. Response options range from 6 (best case) to 0 (worst case). Total scores for treatment satisfaction range from 0-36. Higher scores indicate higher satisfaction. Study GMAJ was terminated after enrolling 38 participants. Given the small sample size overall and per treatment arm, numerical summaries and statistical comparisons are not appropriate and may be scientifically/clinically misleading; therefore, this outcome measure was not analyzed.
Time Frame: Baseline, 12 weeks, 16 weeks
Population: Quality of life data were not analyzed due to insufficient sample size.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LY2599506 | Glyburide
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change From Baseline in the Adult Low Blood Sugar Survey (LBSS-33 Item Scale) at 12 Weeks and 16 Weeks
Description: Assesses 2 hypoglycemia domains, with each item score from 0 (never engages in behavior) to 4 (always engages in behavior): Behavioral (15 items; range 0-60) and Worry about hypoglycemia (18 items; range 0-72). Total score is the sum of both domains (range 0-132). Higher scores indicate greater negative impact. Study GMAJ was terminated after enrolling 38 participants. Given the small sample size overall, and per treatment arm, numerical summaries and statistical comparisons are not appropriate and may be scientifically/clinically misleading. As a result, this outcome measure was not analyzed.
Time Frame: Baseline, 12 weeks, 16 weeks
Population: Quality of life data were not analyzed due to insufficient sample size.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LY2599506 | Glyburide
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Changes From Baseline in the Diabetes Symptoms Checklist-Revised (DSC-R) at 12 Weeks and 16 Weeks
Description: Comprise 6 subscales (34 items). Each item score: 1 (not troublesome) to 5 (extremely troublesome) and transformed to 0-4 scale. Subscale score=sum of item scale in each subscale/total number of items. Global score=sum of scores by dimension. All scores standardized (0-100). Higher scores=greater symptom burden. Study GMAJ was terminated after enrolling 38 participants. Given the small sample size overall and per treatment arm, numerical summaries and statistical comparisons are not appropriate and may be scientifically/clinically misleading; therefore, this outcome measure was not analyzed.
Time Frame: Baseline, 12 weeks, 16 weeks
Population: Quality of life data were not analyzed due to insufficient sample size.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LY2599506 | Glyburide
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change From Baseline in the Perceptions About Medications - Diabetes (PAM-D) Questionnaire at 12 Weeks and 16 Weeks
Description: PAM-D assesses participants' perceptions about their diabetes medications during the past month. Responses ranged from "None of the time," to "All of the time." The sum of all items in the scale equals the scale score, which was linearly transformed to a 0 (least favorable state) to 100 (most favorable state). Study GMAJ was terminated after enrolling 38 participants. Given the small sample size overall and per treatment arm, numerical summaries and statistical comparisons are not appropriate and may be scientifically/clinically misleading; therefore, this outcome measure was not analyzed.
Time Frame: Baseline, 12 weeks, 16 weeks
Population: Quality of life data were not analyzed due to insufficient sample size.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LY2599506 | Glyburide
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at 12 Weeks and 16 Weeks
Description: Change in SBP and DBP following 12 weeks of therapy (Week 12 SBP minus SBP at baseline; Week 12 DBP minus DBP at baseline) and 16 weeks of therapy (Week 16 SBP minus SBP at baseline; Week 16 DBP minus DBP at baseline). Study GMAJ was terminated after enrolling 38 participants. Given the small sample size overall and per treatment arm, numerical summaries and statistical comparisons are not appropriate and may be scientifically/clinically misleading; therefore, this outcome measure is not presented.
Time Frame: Baseline, 12 weeks, 16 weeks
Population: Data were reviewed but are not presented due to insufficient sample size.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | LY2599506 | Glyburide
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Number of Hypoglycemic Episodes During 12-week Treatment Period and 4-week Follow-up Period
Description: Hypoglycemia was defined as any time a participant felt s/he was experiencing a sign or symptom associated with hypoglycemia or had a blood glucose <70 milligrams per deciliter (mg/dL) (3.9 millimoles per liter [mmol/L]) even if it was not associated with signs or symptoms of hypoglycemia. Study GMAJ was terminated after enrolling only 38 participants. Given the small sample size overall and per treatment arm, numerical summaries and statistical comparisons are not appropriate and may be scientifically/clinically misleading; therefore, this outcome measure is not presented.
Time Frame: Baseline through 16 weeks
Population: Data were reviewed but are not presented due to insufficient sample size.
Measure: Number; unit: hypoglycemic episodes
Arm/Group | LY2599506 | Glyburide
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Change From Baseline in Body Weight at 12 Weeks and 16 Weeks
Description: Weight was measured in the fasting state (with the exception of Visit 1) and after emptying the bladder. Participants were instructed to be lightly clothed and without shoes. Study GMAJ was terminated after enrolling 38 participants. Given the small sample size overall and per treatment arm, numerical summaries and statistical comparisons are not appropriate and may be scientifically/clinically misleading; therefore, this outcome measure is not presented.
Time Frame: Baseline, 12 weeks, 16 weeks
Population: Data were reviewed but are not presented due to insufficient sample size.
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | LY2599506 | Glyburide
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Change From Baseline in the Seven-Point Self-Monitored Blood Glucose (7-point SMBG) at 4 Weeks, 12 Weeks, and 16 Weeks
Description: SMBG levels were measured at the following 7 timepoints during the day: fasting prebreakfast, 2 hours post-breakfast, prior to lunch, 2 hours post-lunch, prior to dinner, 2 hours postdinner, and prior to bed. Study GMAJ was terminated after enrolling only 38 participants. Given the small sample size overall and per treatment arm, numerical summaries and statistical comparisons are not appropriate and may be scientifically/clinically misleading; therefore, this outcome measure is not presented.
Time Frame: Baseline, 4 weeks, 12 weeks, 16 weeks
Population: Data were reviewed but are not presented due to insufficient sample size.
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | LY2599506 | Glyburide
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Percentage of Participants With Lipase and Amylase Measurements Above 2-fold Upper Limits of Normal (ULN) During the 12-week Treatment Period
Description: Lipase and amylase concentrations were assessed. Amylase normal limits for males and females are 28-100 units per liter (U/L) (18-50 years), 28-120 U/L (50-60 years), and 28-150 U/L (60-70 years). Normal lipase limits for males and females are 0-100 U/L (18-50 years; 50-60 years) and 0-120 U/L (60-70 years). Study GMAJ was terminated after enrolling only 38 participants. Given the small sample size overall and per treatment arm, numerical summaries and statistical comparisons are not appropriate and may be scientifically/clinically misleading; therefore, this outcome measure is not presented.
Time Frame: Baseline through 12 weeks
Population: Data were reviewed but are not presented due to insufficient sample size.
Measure: Number; unit: percentage of participants
Arm/Group | LY2599506 | Glyburide
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Percentage of Participants With Clinically-Significant Elevations of Alanine Aminotransferase/Serum Glutamate Pyruvate Transaminase (ALT/SGPT) During the 12-week Treatment Period
Description: Clinically significant elevations of ALT/SGPT were considered ≥3 times the upper limit of normal (ULN). The percentage of participants above 2- and 5-fold ULN was not analyzed due to the early termination of the trial. The percentage of participants with ALT 3-fold ULN or higher is presented.
Time Frame: Baseline through 12 weeks
Population: Only randomized participants with a baseline value and at least 1 post-baseline value of the response variable were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | LY2599506 | Glyburide
Number analyzed (Participants) | 16 | 22
percentage of participants | 18.8 | 0

17. Secondary Outcome: Maximum Plasma Concentration (Cmax) at the Steady State for LY2599506
Description: The Cmax value measures the maximum plasma concentration at steady state following administration of doses of LY2599506. Due to the nature of the sparse sampling approach, Cmax was estimated using the posthoc pharmacokinetic (PK) parameters obtained from Population PK (PopPK) modeling. Study GMAJ was terminated after enrolling 38 participants. Given the small sample size overall and per treatment arm, numerical summaries and statistical comparisons are not appropriate and may be scientifically/clinically misleading; therefore, this outcome measure is not presented.
Time Frame: Predose and 2 hours after dosing or predose and 4-12 hours after dosing in weeks 1, 2, 3, and 12
Population: Data were reviewed but are not presented due to the insufficient sample size and sparse sampling approach.
Measure: Mean (Standard Deviation); unit: nanograms per deciliter (ng/dL)
Arm/Group | LY2599506 | Glyburide
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Area Under the Concentration-Time Curve (AUC) at a Dosing Interval (AUCtau) at the Steady State for LY2599506
Description: The AUCtau values measure the area under the plasma concentration time curve at a dosing interval at steady state for LY2599506. Due to the nature of sparse sampling approach taken for the study AUC tau was estimated using the posthoc pharmacokinetic (PK) parameters obtained from Population PK (Pop PK) modeling. Study GMAJ was terminated after enrolling 38 participants. Given the small sample size overall and per treatment arm, numerical summaries and statistical comparisons are not appropriate and may be scientifically/clinically misleading; therefore, this outcome measure was not analyzed.
Time Frame: Predose and 2 hours after dosing or predose and 4-12 hours after dosing in weeks 1, 2, 3, and 12
Population: Data were reviewed but are not presented due to the insufficient sample size and sparse sampling approach.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter times hour
Arm/Group | LY2599506 | Glyburide
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: 30-day Adjusted Rates of Self-reported Hypoglycemic Episodes Overall
Description: Hypoglycemia: any time a participant experienced a sign/symptom associated with hypoglycemia or had blood glucose <70 milligrams per deciliter (mg/dL) (3.9 millimoles per liter [mmol/L]). The 30-day adjusted rate=(total number of episodes between 2 time intervals/number of days between intervals) X 30 days. Study GMAJ was terminated after enrolling 38 participants. Given small sample size overall and per treatment arm, numerical summaries and statistical comparisons are not appropriate and may be scientifically/clinically misleading; therefore, this outcome measure is not presented.
Time Frame: Baseline through 16 weeks
Population: Data were reviewed but are not presented due to insufficient sample size.
Measure: Number; unit: hypoglycemic episodes per 30 days
Arm/Group | LY2599506 | Glyburide
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Change From Baseline in Heart Rate at 12 Weeks and 16 Weeks
Description: Heart rate was measured in heartbeats per minute. Study GMAJ was terminated after enrolling 38 participants. Given the small sample size overall and per treatment arm, numerical summaries and statistical comparisons are not appropriate and may be scientifically/clinically misleading; therefore, this outcome measure is not presented.
Time Frame: Baseline, 12 weeks, 16 weeks
Population: Data were reviewed but are not presented due to the insufficient sample size.
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | LY2599506 | Glyburide
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Mean Morning Dose of LY2599506 During the 12-week Treatment Period
Description: Assigned morning dose, in milligrams (mg), for each participant at each visit. Study GMAJ was terminated after enrolling 38 participants. Given the small sample size overall and per treatment arm, numerical summaries and statistical comparisons are not appropriate and may be scientifically/clinically misleading; therefore, this outcome measure is not presented.
Time Frame: Baseline, 1, 2, 3, 4, 6, 8, 10, 12 weeks.
Population: Data were reviewed but are not presented due to insufficient sample size.
Measure: Mean (Standard Deviation); unit: milligrams (mg)
Arm/Group | LY2599506 | Glyburide
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Mean Afternoon Dose of LY2599506 During the 12-week Treatment Period
Description: Assigned afternoon dose, in milligrams (mg), for each participant at each visit. Study GMAJ was terminated after enrolling 38 participants. Given the small sample size overall and per treatment arm, numerical summaries and statistical comparisons are not appropriate and may be scientifically/clinically misleading; therefore, this outcome measure is not presented.
Time Frame: Baseline, 1, 2, 3, 4, 6, 8, 10, 12 weeks.
Population: Data were reviewed but are not presented due to insufficient sample size.
Measure: Mean (Standard Deviation); unit: milligrams (mg)
Arm/Group | LY2599506 | Glyburide
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Percentage of Participants Requiring Dose Adjustments During the 12-week Treatment Period
Description: Percentage of participants who required dose adjustments at the discretion of the investigator for participants with persistent blood glucose<70 milligrams per deciliter (mg/dL). Study GMAJ was terminated after enrolling 38 participants. Given the small sample size overall and per treatment arm, numerical summaries and statistical comparisons are not appropriate and may be scientifically/clinically misleading; therefore, this outcome measure is not presented.
Time Frame: Baseline through 12 weeks
Population: Data were reviewed but are not presented due to insufficient sample size.
Measure: Number; unit: percentage of participants
Arm/Group | LY2599506 | Glyburide
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: Mean Total Daily Dose of LY2599506 During the 12-week Treatment Period
Description: The average total daily dose (sum of assigned morning and afternoon doses), in milligrams (mg), at each visit. Study GMAJ was terminated after enrolling 38 participants. Given the small sample size overall and per treatment arm, numerical summaries and statistical comparisons are not appropriate and may be scientifically/clinically misleading; therefore, this outcome measure is not presented.
Time Frame: Baseline through 12 weeks.
Population: No participants had data analyzed due to insufficient sample size.
Measure: Mean (Standard Deviation); unit: milligrams (mg)
Arm/Group | LY2599506 | Glyburide
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | LY2599506 | Glyburide
Serious Adverse Events (participants affected / at risk) | 1/16 | 0/22
Other Adverse Events (participants affected / at risk) | 5/16 | 5/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2599506 (N=16) | Glyburide (N=22)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2599506 (N=16) | Glyburide (N=22)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Infectious mononucleosis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Since Study GMAJ was terminated after enrolling only 38 participants with just 1 participant completing 12 weeks of treatment, only disposition, demographics, and safety data are reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less